CLINICAL TRIAL: NCT07199361
Title: Uncovering the Mechanism of Pain Relief by Peripheral Transcutaneous Magnetic Stimulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Collaborators: Baptist Health South Florida (Other)
Responsible Party: Principal Investigator, Dr. Saurabh Aggarwal, Associate Professor, Florida International University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB-25-0065
Record Dates: First submitted 2025-09-21; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Post-Surgical Pain, Chronic; Post-traumatic Pain, Chronic
Keywords: Peripheral Transcutaneous Magnetic Stimulation; Post-Traumatic and Post-Surgical Chronic Pain
MeSH Terms: conditions — Pain, Postoperative; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Intervention Model Description: The study is a "pre vs. post" pTMS therapy, a one-group pretest-posttest study model. In this model, all the study participants will undergo pTMS for 4 consecutive days, and the changes in the mediators of chronic pain in plasma, serum, and peripheral immune cells will be measured in therapy responders and non-responders before pTMS and again after pTMS. The goal is to see if the intervention caused a change in the outcome within that same group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Post-traumatic or post-surgical chronic pain (Experimental): Arm Description: 50 Participants with post-surgical or post-traumatic chronic pain below the neck will be administered peripheral transcutaneous magnetic stimulation at the site of pain for 13 minutes for 4 consecutive days. Participants will be male or female between the ages of 19 and 80 years.
  Interventions: Device: Peripheral Transcutaneous Magnetic Stimulation from MagVenture

INTERVENTIONS:
Device: Peripheral Transcutaneous Magnetic Stimulation from MagVenture — MagVenture Pain Therapy System: It is an FDA-cleared magnetic stimulator system that provides brief and focused magnetic pulses to non-invasively stimulate peripheral nerves and provide relief of chronic intractable, post-traumatic, and post-surgical pain for patients 18 years or older. It is a relatively new technique in the US for pain relief in the clinical setting and thus not very widespread yet. Evidence shows Magnetic Peripheral Nerve Stimulation to have a promising average pain relief of up to 87%*. Using magnetic pulses, MagVenture Pain Therapy engages sensory, pain, and motor fibers mechanistically to recondition the central nervous system by eliminating noxious pain signals to the brain, reducing chronic neuropathic pain for responsive patients.
  *Bedder M, Parker L.: Magnetic Peripheral Nerve Stimulation (mPNS) for Chronic Pain, 2023

SUMMARY:
This research aims to uncover the Mechanisms of pain relief through the FDA-cleared peripheral transcutaneous magnetic stimulation (pTMS) device by MagVenture. 50 people with chronic pain (post-surgical or post-traumatic) will be identified and recruited. The eligibility for participation in the study will be evaluated by a series of pain and mental health questionnaires followed by quantitative sensory testing (QST) to assess response to noxious heat, cold, and pressure stimuli. Blood will be drawn to isolate plasma, serum, and leukocytes. Participants will then undergo pTMS at the site of pain for four consecutive days. At the end of the therapy, pain testing will be done again, followed by blood withdrawal to assess the changes in plasma and leukocyte levels of mediators of pain. It is anticipated that pTMS will increase mediators of pain relief and reduce inflammatory mediators. Risks: It is possible that a few participants may not respond to pTMS therapy. However, plasma analysis of mediators of pain may help stratify these participants into responders vs. non-responders. Risks associated with the study are minimal and mainly involve discomfort associated with pain testing. The importance of knowledge gained includes understanding pain relief mechanisms by medical devices such as pTMS, which will result in better pain management.

DETAILED DESCRIPTION:
Chronic pain (pain lasting ≥3 months) is a debilitating condition associated with depression, dementia, increased risk of suicide, decreased productivity, and substance abuse. Opioids continue to be a crucial part of pain management. However, the misuse of prescription opioids has led to a shift towards injectable opioids such as heroin, with nearly 80% of new heroin users reporting prior use of prescription opioids. Further, co-morbid substance abuse can exacerbate pain symptoms despite pharmaceutical treatment, revealing the limitations of current pain management strategies. Due to tolerance, people with a history of opioid dependence often need higher doses of opioids to treat acute pain and long-term opioid use paradoxically worsens chronic pain. From a public health perspective, there is an increased chance of transmitting and acquiring hepatitis B and C due to opioid use-related engagement in risky behaviors. Moreover, the economic burden of untreated pain in the US is estimated to be more than $100 billion per year. Therefore, there is an urgent need to develop novel therapeutic strategies and reduce reliance on opioids.

Peripheral Transcutaneous Magnetic Stimulation (pTMS) is a non-invasive method of relieving pain by stimulating the target area with magnetic pulses. The magnetic field pulse passing into the body induces a voltage difference between any two points, which creates an electric field and causes electrons to flow between these two points. The magnetic field can penetrate deep tissue, such as spinal nerve roots or muscles. No mechanical contact is necessary, making pTMS applicable to patients with extreme hypersensitivity or allodynia to skin touch. pTMS is FDA-cleared for post-traumatic and post-surgical chronic pain. However, to date, no clear evidence has emerged about pTMS's potential mechanism of pain relief, which has moderated its applicability and acceptability.

The study will require recruiting patients over the phone, followed by an on-site visit, which includes patient interaction, blood collection, pain study, performing pTMS therapy at the site of pain, and patient monitoring. Three more on-site visits on consecutive days will include pTMS therapy. The last (fourth) visit will include specimen collection and a pain study. The first and the fourth visits will take 2.5 hours, while the second and the third visits will require 30 minutes. The participants will be followed over the phone every 30 days till the completion of the study to inquire about their wellness.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of chronic peripheral pain secondary to trauma or surgery. Age 19 - 80; the lower end of this age range was chosen to capture young adults with pain, and participants over 80 years are increasingly likely to meet one or more exclusion criteria.

Currently receiving pain medication Chronic pain must self-report peripheral pain, more than once per week, for at least three consecutive months

Exclusion Criteria:

* Implanted Electronic Devices and / or Conductive Objects in or near the head: Patients who have an implanted device that is activated or controlled in any way by physiological signals (examples: deep brain stimulators, cochlear implants, and vagus nerve stimulators).

Non-Removable Metallic Objects near the coil: Patients who have conductive, ferromagnetic, or other magnetic-sensitive metals implanted in their head or within 30 cm of the treatment coil (examples: cochlear implants, implanted electrodes/stimulators, aneurysm clips or coils, stents, and bullet fragments). F NOTE: Standard amalgam dental fillings are not affected by the magnetic field and are acceptable in patients.

Active microbial infections may alter the quantity or quality of blood inflammatory cells such as monocytes and neutrophils.

Positive Urine Drug test: (COC/AMP/OPI/mAMP/PCP/BAR/BZO/MTD/MDMA/OXY/PPX/BUP/TCA) Use of any medication other than pain medications. However, participants will not be excluded or asked to withdraw from medications used for pain management since temporary withdrawal from these medications could affect pain measures (exceptions will be therapies such as methadone or buprenorphine used to treat opioid addiction). Only those who have been stable on these medications for at least 60 days will be included. All patient medications used for at least 60 days prior to participation will be recorded and controlled in statistical analyses as needed.

Systemic rheumatic disease (e.g., rheumatoid arthritis, systemic lupus erythematosus). These rheumatologic conditions will be excluded due to their autoimmune characteristic.

Cachexia (wasting syndrome) and severe frailty as determined by the Groningen Frailty Index (score >4). This exclusion is in place to protect against the stress of experimental pain testing.

Uncontrolled hypertension (i.e. SBP/DBP of >140/90) or cardiovascular or peripheral arterial disease. These exclusions are in place primarily for safety reasons because the cold pressor task represents a cardiovascular challenge. However, uncontrolled hypertension can also affect pain perception, which is another reason for excluding these individuals.

Poorly controlled diabetes (HbA1c > 8%) for both safety reasons and because diabetic neuropathy could alter pain perception.

Neurological disease (e.g. Parkinson's, multiple sclerosis). Serious psychiatric disorder requiring hospitalization within the past 12 months or characterized by active suicidal ideation. Any participant deemed to be actively suicidal upon study screening will be escorted to the emergency room and evaluated by the Psychiatry Service.

A diminished cognitive function that would interfere with the understanding of study procedures. The Mini-Mental Status Exam (MMSE) will be administered to ensure that participants are free of cognitive impairment that would compromise study participation. MMSE <18 will be excluded.

Pregnancy

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-03-24 (Actual); Primary Completion 2028-01-25 (Estimated); Study Completion 2028-02-25 (Estimated)

PRIMARY OUTCOMES:
Pressure Pain Assessment | 1. On Day 1 (Baseline) 2. On Day 4 (post therapy)
  Pressure Pain Threshold. A handheld probe (Algomed, Medoc) with a small (less than ½ inch wide) rubber tip will be used to apply pressure to the participant's forearm and shoulder. The pressure will slowly increase, and the participant will be asked to click a button when they first feel pain as a result of the pressure stimulation. The pressure will be removed as soon as the participant presses this button. This particular algometer will be used because it provides the examiner with visual feedback to maintain a consistent application rate, which is critical for maintaining high inter-examiner reliability. To assess the pressure pain threshold, the examiner will apply a constant rate of pressure, and the participant will be instructed to press a button when the sensation first becomes painful, at which time the device records the pressure in kilopascals. Higher kilopascals would suggest less pressure pain.
Thermal (Heat) pain | 1. On day 1 (Baseline) 2. On day 4 (Post therapy)
  Thermal (Heat) (Threshold, pain, and tolerance) will be assessed using TSA2 Air device from Medoc:
  A slowly increasing heat stimulus that the participant can terminate by pressing a button when it becomes painful or intolerable. The participant would press the button when they first feel warm (threshold), pain, or can no longer tolerate the heat.
  Lower heat indices indicate higher thermal sensitivity.
Thermal (Cold) Pain | 1. On day 1 (Baseline) 2. On day 4 (Post therapy)
  Thermal (Cold) (Threshold, pain, and tolerance) will be assessed using TSA2 Air device from Medoc: A slowly decreasing cold stimulus that the participant can terminate by pressing a button when it becomes painful or intolerable. The participant would press the button when they first feel cold (threshold), pain, or can no longer tolerate the cold. Higher cold indices indicate higher thermal sensitivity.
Temporal Heat Summation | 1. On day 1 (Baseline) 2. On Day 4 (Post therapy)
  Temporal heat summation will be measured using TSA2 Air device. A series of 5 brief heat pulses (about 2 seconds in duration) will be given, and the participant will be asked to rate how painful each heat pulse feels on a scale from 0 to 100. These heat pulses will be repeated at different temperatures (44° C, 46° C, and 48° C). The participant can stop the procedures at any time so that they do not experience unacceptable pain.
  Greater pain ratings indicate more pain
Conditioned Pain Modulation | 1. On day 1 (Baseline) 2. On day 4 (Post Therapy)
  Conditioned pain modulation (CPM) will be tested by TSA2 Air Device. The standard thermode will be placed on the left hand, and the heat pain rating will be assessed at 46 degrees. Then the right hand will be immersed in cold water for 30 seconds. The Heat pain test will be performed again on the left hand to assess Pain modulation.
  A normal response would indicate a decrease in heat pain on the left hand after immersing the right hand in cold water.

SECONDARY OUTCOMES:
McGill Pain Questionnaire-Short Form | 1. On day 1 (Baseline) 2. On day 4 (Post therapy)
  Description: 15 descriptors (11 sensory; 4 affective) using an intensity scale ranging from 0-3 on the pain scale (0 = no pain, 1 = mild pain, 2 = moderate pain, or 3 = severe pain) A higher number indicates more pain
Brief Pain Inventory | 1. On day 1 (Baseline) 2. On day 4 (Post therapy)
  A set of 4 Pain Questionnaire:
  Worst pain in last 24 hours: (1-10) Least pain in last 24 hours (1-10) Pain on average (1-10) Pain right now (1-10) Total possible score: 40 A higher number indicates more pain
Present Pain Index | 1. On day 1 (Baseline) 2. On day 4 (Post therapy)
  A pain score of current pain on the scale of 0-5 A higher number indicates more pain
Visual Analogue scale | 1. On day 1 (Baseline) 2. On day 4 (Post therapy)
  A visual pain scale of 1-100 A higher number indicates more pain
PHQ-9 | 1. On day 1 (Baseline) 2. On day 4 (Post therapy)
  Patient Health Questionnaire (depression screening) Scores : 0-27 A higher number indicates greater depression
GAD-7 | 1. On day 1 (Baseline) 2. On day 4 (Post therapy)
  General Anxiety Disorder 7 items scored between 0-3. Score: 0-21 A higher number indicates more anxiety
Vascular Reactivity Index (VRI) | 1. On day 1 (Baseline) 2. On day 4 (Post therapy)
  A vascular function test using the Vendys Endothelix device Measures Vascular function Score: 0-3 (VRI) The higher the number, the better the vascular function.
Measuring Endogenous Opioids in Plasma | 1. On day 1 (Baseline) 2. On day 4 (Post therapy)
  20 ml of blood will be drawn to isolate plasma and peripheral leukocytes in pg/ml. Lower endogenous opioids indicate more pain.
Measuring Inflammatory cytokines in Plasma | 1. On Day 1 (Baseline) 2. On Day 4 (Post Therapy)
  A 20 ml blood sample will be collected, and plasma cytokines will be measured in mg/ml.
  Higher plasma cytokines indicate more pain
Measuring endogenous opioids in peripheral immune cells. | 1. On day 1 (Baseline) 2. On day 4 (Post Therapy)
  A 20 ml blood sample will be collected, and endogenous opioids will be measured in pg/mg protein.
  Lower endogenous opioids would indicate more pain

CONTACTS AND LOCATIONS:
Overall Officials: Saurabh Aggarwal, MD., PhD, Principal Investigator — Florida International University; Patricia Junquera, MD, Principal Investigator — Florida International University and Baptist Health South Florida; Eduardo Icaza, MD, Principal Investigator — Baptist Health South Florida
Locations (1):
- Ambulatory Care Center, Florida International University, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in Chronic Pain. Data or samples shared will be coded, with no PHI included. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party
Supporting Information: CSR
Time Frame: Data requests can be submitted starting 9 months after article publication, and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA).